CLINICAL TRIAL: NCT00497861
Title: Comparison of Mechanical Force, Manually Assisted Activator Manipulation Versus Manual Side Posture Manipulation in Patients With Low Back Pain: a Randomized Pilot Study
Brief Title: Comparison of Activator Manipulation Versus Manual Side Posture Manipulation in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Chiropractic College (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPMFMA1
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2007-07-09 (Estimated); Status verified 2007-04

CONDITIONS: Back Pain
Keywords: Low back pain; Chiropractic; Spinal manipulation; Activator Methods Chiropractic Technique
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Activator Methods Chiropractic Technique

SUMMARY:
This study compared the treatment effect of Activator Methods Chiropractic Technique (AMCT) and manual Diversified type spinal manipulative therapy in a sample of patients with acute and sub-acute low back pain.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects of (MFMA) Activator instrument adjusting to manual side posture (HVL) adjustments in patients with acute low back pain.

Primary outcomes measured include pain measurement with a VAS scale, the use of the Oswestry pain scale questionnaire, and the Bournemouth back pain scale questionnaire.

An additional aim of this study is to evaluate feasibility of recruitment, data collection, and other procedures which can lead to additional studies with larger number of subjects including a control group.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18 years or older;
2. Having current acute or sub-acute low back pain defined as pain that has not lasted more than 16 weeks;
3. Minimum score of 30mm on a 100mm visual analog pain scale.

Exclusion Criteria:

Exclusion criteria consisted of the following:

1. Have any of six possible un underlying causes of low back symptoms in their history (spinal osteomyletisosteomyelitis, spinal fracture, herniated disc, ankylosing spondylitis, cauda equina syndrome, or cancer, excluding nonmalignant skin cancer);
2. Have undergone surgery involving the low back; (
3. Have received workers'compensation benefits within the preceding year or were potentially involved in litigation relating to back problems;
4. Pregnancy, because of possible need for exposure to diagnostic x-rays;
5. Have participated as a subject in research previously at the trial clinic site;
6. Have received spinal manipulation within the preceding 3 months or on more than three occasions during the preceding year.
7. Subjects with sciatica were excluded if they had any one of the following:

   * Ankle dorsiflexion / plantar flexion weakness;
   * Great toe extensor weakness;
   * Absence of knee or ankle reflexes;
   * Loss of light touch sensation in the medial, dorsal, and lateral aspects of the foot;
   * Ipsilateral straight-leg-raising test (positive result: leg pain at <60°);
   * Crossed straight-leg-raising test (positive result: reproduction of contralateral pain).

   These six neurologic tests allow detection of most clinically significant nerve root compromises resulting from L4-L5 or L5-S1 disc herniations, which together make up more than 90% of all clinically significant radiculopathies attributable to lumbar disc herniations (21-25). Because approximately 12% of ambulatory patients with back pain h
8. Have symptoms of sciatica or leg pain without neurologic compromise related to lumbar disc herniation,[5] investigators attempted to include such subjects in the trial.

The criteria described above were intended to minimize the likelihood of including subjects with a lumbar disc herniation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-12; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Revised Oswestry | December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Pfefer, D.C., R.N., Principal Investigator — Cleveland Chiropractic College
Locations (1):
- Cleveland Chiropractic College, Kansas City, Missouri, United States